CLINICAL TRIAL: NCT02084654
Title: Randomized Trial Investigating Exenatide for Diabetes Prevention in Obese, Insulin-Resistant Individuals With Prediabetes
Brief Title: Exenatide and Weight Loss for Diabetes Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 9946
Record Dates: First submitted 2013-12-02; First posted 2014-03-12 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Pre Diabetes; Insulin Resistance
Keywords: prediabetes; exenatide; weight loss; insulin resistance; acute insulin response; insulin secretion
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Prediabetic State; Weight Loss | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- exenatide 5 and 10 mcg 2 times a day (Active Comparator): Exenatide in addition to weight loss. Starting dose 5 mcg titrate to 10 mcg
  Interventions: Drug: Exenatide 5 and 10 mcg 2 times a day
- placebo (Placebo Comparator): placebo in addition to weight loss
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Exenatide 5 and 10 mcg 2 times a day
  Other Names: Byetta
  Arms: exenatide 5 and 10 mcg 2 times a day
Drug: placebo
  Arms: placebo

SUMMARY:
Exenatide, a GLP-1 agonist approved for lowering blood glucose concentrations in patients with type 2 diabetes, has been associated with restoration of the first-phase insulin response when administered intravenously to patients with type 2 diabetes. In longer clinical trials, it is associated with progressive decreases in body weight, and improvement in the dyslipidemia that characterizes insulin resistance, although insulin resistance was not quantified. The investigators will seek to determine whether exenatide would have similar effects in individuals who were not diabetic. in particular, the drug effect on beta cell function and insulin sensitivity would be subject to less confounding by changes in blood glucose in the prediabetic population, allowing for clearer evaluation of the physiological effects of the drug on these metabolic endpoints. The investigators will compare 2 groups of prediabetic insulin resistant individuals, all on a weight loss diet and one group on exenatide and the other on placebo. The investigators will evaluate restoration of first phase insulin response, potential glucose lowering effects, including both reversal of prediabetes and hypoglycemia, and improvement in insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men and women, BMI 27-37kgm2, Fasting plasma glucose = or > 100 mg/dL and = or < 99 125m g/dl or a 2 hour post OGTT = > 140 mg/dl or = or < 199 mg/dl

Exclusion Criteria:

* Diabetes, Active cardiac, kidney, liver, pulmonary, or other major organ diseases are cause for exclusion. Other exclusionary criteria include: use of corticosteroids, diet medications, antipsychotic medications, history of eating disorder, history of bariatric surgery, active malignancy, recent weight change of more than 2%, inability to attend follow-up visits, excessive alcohol use, investigator's discretion that it is not in patient's best interest

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-11; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
First-phase insulin response | 7 months
  measured using ivgtt

SECONDARY OUTCOMES:
glucose lowering effect | 8 months
  measured by fasting and 2 hr plasma glucose during OGTT

OTHER OUTCOMES:
insulin-mediated glucose uptake (insulin sensitivity) | 8 months
  This is measured by the SSPG, or modified insulin-suppression test. it is a "gold standard" measurement of insulin-mediated glucose uptake, and is precise and quantitative.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MS, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No